CLINICAL TRIAL: NCT06084585
Title: A Three Arms, Randomized, Double-blind Controlled Trial of the Efficacy of Amway Uric Acid Lowering Product on Hyperuricemia
Brief Title: The Efficacy of Amway Uric Acid Lowering Product on Hyperuricemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amway (China) R&D Center (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 22-RB-07-AY-001
Record Dates: First submitted 2023-10-10; First posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Hyperuricemia
Keywords: Uric Acid; Amway
MeSH Terms: conditions — Hyperuricemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Study Product A (High-dose 2X) (Active Comparator): Amway uric acid lowering product: 5g/sachet, containing the following active ingredients:
  * Celery seed (functional raw material)
  * Dasiphora mandshurica (functional raw material)
  * Cichorium intybus L. (functional raw material)
  * Lotus leaf (functional raw material)
  * Tart cherry (functional raw material)
  * γ-cyclodextrin
  * Erythritol
  * Silicon dioxide
  * Resistant dextrin
  * Black tea essence
  Interventions: Dietary Supplement: Study Product A (High-dose 2X)
- Study Product B (Low-dose X) (Active Comparator): Amway uric acid lowering product: 5g/sachet, containing the following active ingredients:
  * Celery seed (functional raw material)
  * Dasiphora mandshurica (functional raw material)
  * Cichorium intybus L. (functional raw material)
  * Lotus leaf (functional raw material)
  * Tart cherry (functional raw material)
  * γ-cyclodextrin
  * Erythritol
  * Silicon dioxide
  * Resistant dextrin
  * Black tea essence
  Interventions: Dietary Supplement: Study Product B (Low-dose X)
- Placebo (Placebo Comparator): Placebo product: 5g/sachet, containing the following active ingredients:
  * Maltodextrin
  * Pigment
  * Erythritol
  * Bitters
  * Essence of flavor
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Study Product A (High-dose 2X) — participants in this arm will consume 1 sachet of this product with 200ml water per time, once a day after meal, for 3 months
  Arms: Study Product A (High-dose 2X)
Dietary Supplement: Study Product B (Low-dose X) — participants in this arm will consume 1 sachet of this product with 200ml water per time, once a day after meal, for 3 months
  Arms: Study Product B (Low-dose X)
Dietary Supplement: Placebo — participants in this arm will consume 1 sachet of this product with 200ml water per time, once a day after meal, for 3 months
  Arms: Placebo

SUMMARY:
The goal of this three arms, randomized, double-blind controlled interventional study is to evaluate the efficacy of Amway uric acid lowering product improving hyperuricemia in patients aged 18 and 65 years old. The main question it aims to answer is:

- whether the serum uric acid level of patients with hyperuricemia could be significantly lowered after 3 months intervention with Amway uric acid lowering product

180 eligible participants will be enrolled in one study site and randomized to three study groups (two product group and one placebo group), who will consume the assigned products for 3 months and be arranged to 3 site visits. All relevant clinical data will be captured and recorded into CTMS (Clinical Trial Management System) for statistical analysis and reporting.

Researchers will compare the three study groups to conclude how Amway uric acid lowering product will improve hyperuricemia.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged between 18 and 65 years old (mostly above 35 years old), including male and female and the ratio of male to female is not limited;
* Patients with hyperuricemia: meet the diagnostic criteria set out in the "Chinese Guidelines for Diagnosis and Treatment of Hyperuricemia and Gout (2019)", and fasting blood uric acid level exceeds 420 μmol/L twice on different days. Further classification using the Janssens Gout Diagnostic scale included asymptomatic hyperuricemia (that is, never had a gout attack) and patients with a history of gout, with a ratio of about 1:1;
* Participants agree not to take any drugs, supplements, or performance enhancers during the study, or they will be eliminated
* Participants understand the test procedure, read, and sign an appropriate Informed Consent Form indicating their willingness to participate.

Exclusion Criteria:

* Secondary gout caused by kidney disease, blood disease, drug use, tumor radiotherapy and chemotherapy;
* Subjects who are using drugs during gout attacks;
* Malignant diseases: patients with severe lung, cardiovascular, blood and hematopoietic system, central nervous system or other system diseases, as well as tumor patients;
* Severe obesity (BMI>32kg/m2);
* Abnormal liver and kidney function: abnormal level of alanine aminotransferase or aspartate aminotransferase; Serum creatinine was higher than the upper limit of the normal range;
* Allergic to the test drug or weak or allergic;
* Pregnant or lactating women or those who have pregnancy plans; Sex hormone replacement therapy and oral contraception in the past 3 months;
* Subjects who have participated in other research projects within three months;
* Subjects that other researchers considered should be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-10-23 (Estimated); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-03-15 (Estimated)

PRIMARY OUTCOMES:
Change of Serum Uric Acid Level | baseline, and 12 weeks
  Change of Serum Uric Acid Level from baseline to 12 weeks, in unit of μmol/L, diagnosed as hyperuricemia if the level exceeds 420umol/L twice on different days

SECONDARY OUTCOMES:
Change of Serum Uric Acid Level | baseline, and 6 weeks
  Change of Serum Uric Acid Level from baseline to 6 weeks, in unit of μmol/L, diagnosed as hyperuricemia if the level exceeds 420umol/L twice on different days
Fractional Excretion of Uric Acid (FEUA) | baseline, 6 weeks, and 12 weeks
  Fractional Excretion of Uric Acid (FEUA), defined as the percentage of urate filtered by glomeruli that is excreted in urine, normal range 7~12%. A FEUA value less than 7% considered low, indicating decreased renal excretion of uric acid. A FEUA value above 12% is considered high, suggesting increased renal excretion of uric acid.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Cao, MD, Principal Investigator — Jinhua Wenrong Hospital
Locations (1):
- Charlie Zhang, Jinhua, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dehlin M, Jacobsson L, Roddy E. Global epidemiology of gout: prevalence, incidence, treatment patterns and risk factors. Nat Rev Rheumatol. 2020 Jul;16(7):380-390. doi: 10.1038/s41584-020-0441-1. Epub 2020 Jun 15. PMID 32541923
- [Background] Choi HK, Mount DB, Reginato AM; American College of Physicians; American Physiological Society. Pathogenesis of gout. Ann Intern Med. 2005 Oct 4;143(7):499-516. doi: 10.7326/0003-4819-143-7-200510040-00009. No abstract available. PMID 16204163
- [Background] Zhang M, Zhu X, Wu J, Huang Z, Zhao Z, Zhang X, Xue Y, Wan W, Li C, Zhang W, Wang L, Zhou M, Zou H, Wang L. Prevalence of Hyperuricemia Among Chinese Adults: Findings From Two Nationally Representative Cross-Sectional Surveys in 2015-16 and 2018-19. Front Immunol. 2022 Feb 7;12:791983. doi: 10.3389/fimmu.2021.791983. eCollection 2021. PMID 35197964
- [Background] Li L, Zhang Y, Zeng C. Update on the epidemiology, genetics, and therapeutic options of hyperuricemia. Am J Transl Res. 2020 Jul 15;12(7):3167-3181. eCollection 2020. PMID 32774692
- [Background] Liu N, Wang Y, Yang M, Bian W, Zeng L, Yin S, Xiong Z, Hu Y, Wang S, Meng B, Sun J, Yang X. New Rice-Derived Short Peptide Potently Alleviated Hyperuricemia Induced by Potassium Oxonate in Rats. J Agric Food Chem. 2019 Jan 9;67(1):220-228. doi: 10.1021/acs.jafc.8b05879. Epub 2018 Dec 28. PMID 30562028
- [Background] Gliozzi M, Malara N, Muscoli S, Mollace V. The treatment of hyperuricemia. Int J Cardiol. 2016 Jun 15;213:23-7. doi: 10.1016/j.ijcard.2015.08.087. Epub 2015 Aug 8. PMID 26320372
- [Background] Jiang LL, Gong X, Ji MY, Wang CC, Wang JH, Li MH. Bioactive Compounds from Plant-Based Functional Foods: A Promising Choice for the Prevention and Management of Hyperuricemia. Foods. 2020 Jul 23;9(8):973. doi: 10.3390/foods9080973. PMID 32717824
- [Background] Yang B, Xin M, Liang S, Xu X, Cai T, Dong L, Wang C, Wang M, Cui Y, Song X, Sun J, Sun W. New insight into the management of renal excretion and hyperuricemia: Potential therapeutic strategies with natural bioactive compounds. Front Pharmacol. 2022 Nov 22;13:1026246. doi: 10.3389/fphar.2022.1026246. eCollection 2022. PMID 36483739
- [Background] Li S, Li L, Yan H, Jiang X, Hu W, Han N, Wang D. Anti-gouty arthritis and anti-hyperuricemia properties of celery seed extracts in rodent models. Mol Med Rep. 2019 Nov;20(5):4623-4633. doi: 10.3892/mmr.2019.10708. Epub 2019 Sep 26. PMID 31702020
- [Background] Wang Y, Lin Z, Zhang B, Nie A, Bian M. Cichorium intybus L. promotes intestinal uric acid excretion by modulating ABCG2 in experimental hyperuricemia. Nutr Metab (Lond). 2017 Jun 13;14:38. doi: 10.1186/s12986-017-0190-6. eCollection 2017. PMID 28630638
- [Background] Wang Y, Lin Z, Zhang B, Jiang Z, Guo F, Yang T. Cichorium intybus L. Extract Suppresses Experimental Gout by Inhibiting the NF-kappaB and NLRP3 Signaling Pathways. Int J Mol Sci. 2019 Oct 4;20(19):4921. doi: 10.3390/ijms20194921. PMID 31590257
- [Background] Wang MX, Liu YL, Yang Y, Zhang DM, Kong LD. Nuciferine restores potassium oxonate-induced hyperuricemia and kidney inflammation in mice. Eur J Pharmacol. 2015 Jan 15;747:59-70. doi: 10.1016/j.ejphar.2014.11.035. Epub 2014 Dec 8. PMID 25499818
- [Background] Cheng-Yuan W, Jian-Gang D. Research progress on the prevention and treatment of hyperuricemia by medicinal and edible plants and its bioactive components. Front Nutr. 2023 Jun 12;10:1186161. doi: 10.3389/fnut.2023.1186161. eCollection 2023. PMID 37377486
- [Background] Li R, Tan Y, Li Y, Zhu X, Tang X, Zhang L, Chen J. Effects of Tart Cherry Powder on Serum Uric Acid in Hyperuricemia Rat Model. Evid Based Complement Alternat Med. 2020 Jul 22;2020:1454305. doi: 10.1155/2020/1454305. eCollection 2020. PMID 32774405
- [Background] Chen PE, Liu CY, Chien WH, Chien CW, Tung TH. Effectiveness of Cherries in Reducing Uric Acid and Gout: A Systematic Review. Evid Based Complement Alternat Med. 2019 Dec 4;2019:9896757. doi: 10.1155/2019/9896757. eCollection 2019. PMID 31885677